CLINICAL TRIAL: NCT04953741
Title: A Comparative Study on the Efficacy of Different Stepping-down Therapy for Childhood Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20202053-F-1
Record Dates: First submitted 2021-06-11; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2020-09

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Stop Fluticasone propionate Inhaled Aerosol Firstly (Active Comparator): Reduced dose Fluticasone propionate Inhaled Aerosol 125 ug once a day and continuation of montelukast once a day，and then stopped Fluticasone propionate Inhaled Aerosol and continuation of montelukast once a day
  Interventions: Drug: Fluticasone propionate inhaled aerosol
- Stop Montelukast Secondly (Active Comparator): Reduced dose Fluticasone propionate Inhaled Aerosol 125 ug once a day and continuation of montelukast once a day，and then stopped montelukast and continuation of Fluticasone propionate Inhaled Aerosol 125 ug once a day
  Interventions: Drug: Fluticasone propionate inhaled aerosol
- Stop Montelukast Firstly (Active Comparator): stopped montelukast and continuation of Fluticasone propionate Inhaled Aerosol 125 ug twice daily, and then Reduced dose Fluticasone propionate Inhaled Aerosol 125 ug once a day
  Interventions: Drug: Fluticasone propionate inhaled aerosol

INTERVENTIONS:
Drug: Fluticasone propionate inhaled aerosol — The study consists of two stages and include three groups. Three groups include: Reduced dose Fluticasone propionate Inhaled Aerosol 125 ug once a day and continuation of montelukast once a day，and then stopped Fluticasone propionate Inhaled Aerosol and continuation of montelukast once a day; Reduced dose Fluticasone propionate Inhaled Aerosol 125 ug once a day and continuation of montelukast once a day，and then stopped montelukast and continuation of Fluticasone propionate Inhaled Aerosol 125 ug once a day; Stopped montelukast and continuation of Fluticasone propionate Inhaled Aerosol 125 ug twice daily, and then Reduced dose Fluticasone propionate Inhaled Aerosol 125 ug once a day. The scheme of every group is divided into two stages. Only those whose asthma are well controlled at the end of the first phase will be allowed to proceed to the next phase.

SUMMARY:
This study is a 24-week, randomized, parallel group comparative effectiveness study to evaluate the risk of stepping down therapy for patients with well-controlled asthma treated with combination Inhaled corticosteroids (ICS) and Leukotriene receptor antagonist（LTRA).

DETAILED DESCRIPTION:
Asthma guidelines recommend stepping down therapy once asthma is controlled for at least 3 months. Leukotriene receptor antagonist（LTRA). For children with mild persistent asthma, ICS twice a day combined with LTRA can be used for treatment, but there is no consensus on how to reduce drugs in patients with asthma that is well controlled (reducing the dose of ICS or stopping montelukast). We propose a 24-week, randomized, parallel group comparative effectiveness study comparing three approaches in patients with asthma well-controlled for at least three months on combination ICS and LTRA: Halve the dose of ICS firstly and then stop ICS with montelukast only, stop montelukast firstly and then halve the dose of ICS, and halve the dose of ICS firstly and then stop montelukast. Our goal is to compare the rate of treatment failure and determine the optimal treatment strategy. Additional goals include assessing risk factors for step-down failure.

ELIGIBILITY:
Inclusion Criteria:

* age 4-14 years
* patients had mild to moderate persistent asthma. Patients have treated with low-dose inhaled corticosteroids (equivalent to Fluticasone propionate inhaled aerosol 250 ug/ day) combined with Leukotriene receptor antagonist (Montelulast) at least 6 months of and had no symptoms of asthma for nearly 3 months under well asthma control(Asthma Control Test (ACT) score more than or equal to 20).
* patients did not suffer from other acute or chronic diseases that may affect their growth and development

Exclusion Criteria:

* patients with severe persistent asthma or mild persistent asthma failed to be well controlled by low-dose ICS after starting treatment
* suffer from other diseases: Congenital heart disease, chronic infectious disease, protracted diarrhea, congenital airway disease, congenital vascular ring malformation, congenital immune deficiency, tracheal foreign body, bronchial lymph node tuberculosis and gastroesophageal reflux etc.
* patients with poor compliance stop medication or fail to take medication on time.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) score | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
  Change in participant's Asthma Control Test (ACT) score
Number of Participants Who Experienced asthma exacerbation or used oral/intravenous corticosteroids as needed | Baseline (Week 0) to Week 12
  Participants Experienced asthma exacerbation or used oral/intravenous corticosteroids as needed
Number of Participants Who Experienced asthma exacerbation or used oral/intravenous corticosteroids as needed | Baseline (Week 0) to Week 24
  Participants Experienced asthma exacerbation or used oral/intravenous corticosteroids as needed

SECONDARY OUTCOMES:
Fractional exhaled Nitric Oxide, FeNO | Baseline, 12 weeks and 24 weeks
  Change in participant's Fractional exhaled Nitric Oxide
Forced expiratory volume in one second in predicted（FEV1%pred） | Baseline, 12 weeks and 24 weeks
  Change in participant's Forced expiratory volume in one second in predicted
Forced vital capacity in predicted(FVC%pred) | Baseline, 12 weeks and 24 weeks
  Change in participant's Forced vital capacity in predicted
Maximal mid expiratory flow in predicted(MMEF%pred) | Baseline, 12 weeks and 24 weeks
  Change in participant's Maximal mid expiratory flow in predicted
Peak expiratory flow (PEF) | Baseline, 12 weeks and 24 weeks
  Change in participant's Peak expiratory flow

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Xijing Hospital, Xi’an, Shanxi, China

REFERENCES:
- [Result] Bernstein JA, Mansfield L. Step-up and step-down treatments for optimal asthma control in children and adolescents. J Asthma. 2019 Jul;56(7):758-770. doi: 10.1080/02770903.2018.1490752. Epub 2018 Sep 12. PMID 29972079